CLINICAL TRIAL: NCT05625152
Title: Dating of Child Fractures : Chronological Repers From the Radiological Evolution of a Series of Femur Fractures
Acronym: DFE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7955
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-11

CONDITIONS: Fractures in Children
Keywords: Femur Fracture; FRACTURES IN CHILDREN; Pediatric population; Bony Callus
MeSH Terms: conditions — Femoral Fractures; Callosities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although several studies have studied the predictive nature of non-accidental trauma of the different types of fractures and in particular on the femur, the physiological and radiological particularities of the child make it difficult to estimate the age of a fracture and require defining a chronology specific to the specificities of the pediatric population. Some authors have carried out work for the dating of fractures, however the number of cases or the average age of the subjects does not allow a precise estimation of the chronology of evolution of the fractures.

ELIGIBILITY:
Inclusion criteria:

* Child aged 18, cared for in the pediatric orthopedic department of the Strasbourg University Hospitals between January 2007 and December 2020
* Fracture of the femur resulting from orthopedic treatment instituted during a period of hospitalization
* Holders of parental authority who have been informed of the use of their child's data for the purposes of this research and who have not expressed any opposition

Exclusion criteria:

* Patient or legal representative who expressed their opposition to participating in the study
* Fracture of the femur having benefited from a surgical intervention
* Weakening metabolic or bone pathology
* Fracture on pathological focal lesion
* Fractures of the epiphysis or affecting the growth cartilage
* Impossibility of giving informed information to the subject

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child aged 18, cared for in the pediatric orthopedic department of the Strasbourg University Hospitals between January 2007 and December 2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Define retrospectively the chronology of the appearance of periosteal callus, secondary callus and remodeling phenomena from the study of radiographs of the femur | Files analysed retrospectively from January 01, 2007 to December 31, 2020 will be examined
  Evaluation of the time to radiographic appearance of the following stages defined by the number of days elapsed between the date of diagnosis of the fracture and the first radiography taken during follow-up, making it possible to highlight one of these phenomena:
  * The radiographic periosteal reaction (or periosteal callus) defined by an opacity at the periphery of the fracture, corresponding to the first objectifiable calcification of the fracture hematoma and under the periosteum.
  * The secondary bone callus (or osteochondral) defined by a well-defined bone apposition of density close to that of the bone with opacification of the fracture line and union of the fracture site
  * Established remodeling activity when phenomena of axis correction, resorption of initial callus hypertrophy or re-permeabilizatio of the diaphyseal shaft can be demonstrated

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Pédiatrique - CHU de Strasbourg - France, Strasbourg, France